CLINICAL TRIAL: NCT00526500
Title: Effect of Proprioceptive Stimulation With Passive Gait Training on the Cortical Activity in Patients With Impaired Consciousness Due to Severe Brain Injury.
Brief Title: Effect of Passive Gait Training on the Cortical Activity in Patients With Severe Brain Injury.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Natallia Lapitskaya, MD, Hammel Neurorehabilitation and Research Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNRC-AAU-07-1
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Craniocerebral Trauma; Traumatic Brain Injury; Subarachnoid Hemorrhage; Anoxic Brain Injury
Keywords: Severe Traumatic Brain Injury; Subarachnoid Hemorrhage; Anoxic Brain Injury; Passive Gait Training; Tilt Table With Integrated Stepping System; Electroencephalogram; Event Related Potentials
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- P-T (Experimental)
  Interventions: Behavioral: Tilt Table With Integrated Stepping System
- P- SAH (Experimental)
  Interventions: Behavioral: Tilt Table With Integrated Stepping System
- P- A (Experimental)
  Interventions: Behavioral: Tilt Table With Integrated Stepping System
- Control (Experimental)
  Interventions: Behavioral: Tilt Table With Integrated Stepping System

INTERVENTIONS:
Behavioral: Tilt Table With Integrated Stepping System — Passive Gait Training: one session, 20 minutes, table tilted to 70-80 degrees, speed 60 steps per minute.
  Other Names: P-T:patients, traumatic brain injury; P-SAH:patients, subarachnoid hemorrhage; P-A:patients, anoxi; Control: healthy volunteers

SUMMARY:
The aim of this study is to determine effect of proprioceptive stimulation with passive gait training on the cortical activity in patients with severe brain injury, demonstrated as changes in EEG (electroencephalogram)and ERP (Event Related Potentials).

Hypotheses: 1) Proprioceptive stimulation increases EEG-frequency in patients with impaired consciousness due to severe brain injury.

2) Proprioceptive stimulation increases conductivity speed of the cognitive P300-component of ERP in patients with impaired consciousness due to severe brain injury.

DETAILED DESCRIPTION:
Design: Prospective controlled non-randomized study. Materials and methods: 45 patients with severe brain injury and 15 healthy volunteers will be included in this study.

The study design is illustrated below:

1. Baseline measurement of electroencephalography (EEG) and event related potentials (ERP)
2. Gait training in the tilt table with integrated stepping system(20 min).
3. Control measurement of EEG and ERP Effect parameters: se outcome measures. Statistical evaluation: All collected data will be tested with reference to normal distribution. If the data is not distributed normally, then we will use either a logarithmic transformation before we use parametric statistics, or we will use non-parametric statistics for further calculations.

Further analysis of the data will be done with the help of variance analysis with an inter-individually factor as a group (patients vs control persons) and intra-individually factors as: 1) experimental condition (before vs after training), 2) topographic distribution (anterior vs central vs posterior).

Significance level is set to 0.05 for all effect parameters.

ELIGIBILITY:
Inclusion Criteria:

Patient Goup:

1. Severe Brain Injury
2. Ongoing Impaired State of Consciousness (RLAS<4)
3. Stable Vital Functions
4. Written Consent from Relatives/Legal Guardian

Control Group:

1. No History of Neurological Diseases in the Past
2. Age over 18 years
3. Written Consent -

Exclusion Criteria:

Patient and Control Goup:

1. Age older than 80 years
2. Other Neurological Diseases
3. Lack of BAEP
4. Severe Co-morbidity
5. Pregnancy
6. Tilt table contraindications: orthostatic circulatory problems, unstable fractures, severe osteoporosis, sken problems, joint problems, severe asymmetry (major difference in leg length over 2 cm), co-operation problems (psychotic illnesses or neurotic disturbances), adjustment problems (i.e. integrated stepping system cannot be safely adjusted to the patient)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-08; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
EEG:frequency ratios: Alpha versus delta; alpha and beta versus delta and theta; ERP: latency of P300-component. | immediately after the end og the training

SECONDARY OUTCOMES:
EEG: absolute and relative power in every frequency band; median frequency; | immediately after the end of the training

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Kock-Jensen, MD, Study Director — Hammel Neurorehabilitation and Research Centre; Johannes Jakobsen, MD, DMSc, Study Chair — Department of Neurology, Aarhus University; Natallia Lapitskaya, MD, PhD-stud, Principal Investigator — Hammel Neurorehabilitation and Research Centre
Locations (1):
- Hammel Neurorehabilitation and Research Centre, Hammel, Denmark